CLINICAL TRIAL: NCT05310981
Title: A Randomized Pilot Trial of ICanChange, a Mobile Health Intervention to Reduce Cannabis Use in Young Adults With Psychosis
Brief Title: A Cannabis E-intervention for Young Cannabis Users With Early Psychosis (iCC)
Acronym: iCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21.310
Record Dates: First submitted 2022-02-03; First posted 2022-04-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Intervention Model Description: two-arm parallel, open-labelled, pilot randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: CHAMPS and mEIS (Experimental): Brief mobile application-based psychological intervention based on the principles of motivational interviewing (MI) and cognitive behavioural therapy (CBT). This e-intervention will be completed by the participant using a smart phone. There will be up to a maximum of 24 individual sessions (which includes 3 booster sessions) each lasting approximately 10-15 minutes.
  mEIS: iCC will be administered adjunctively to modified EIS (mEIS), which will include all interventions usually provided through EIS except for any specific psychological interventions (MI, CBT, contingency management) for CUD.
  Interventions: Behavioral: iCanChange
- No Intervention: EIS alone (No Intervention): Early intervention services will be offered as per standard of care following EIS for psychosis and CUD guidelines, at participating clinical sites. Any visits and services offered in control arm will be considered 'usual care' and administered either through in-person clinic visits, community visits, phone calls, or video calls. Relevant service information will be collected for study purposes.

INTERVENTIONS:
Behavioral: iCanChange — iCC is a psychological app based intervention that will be delivered in form of up to 24 brief (10-15 minutes) interactive modules developed based on the principles of Motivational Interviewing (MI) and Cognitive Behavioural Therapy (CBT). During the intervention, participants will be offered MI and CBT-based activities (i.e., modules and strategies) aiming at facilitating change in cannabis use. At any point during the intervention, participants can reference modules that had been completed. Due to the frequency of behavioral stage changes in this population (e.g., regression in behavioral stage of change), stage of change will be monitored regularly throughout the intervention. During the follow-up period (i.e., Week 12-24), participants will have continuous access to the smart phone application and all built-in add-ons as described above. During this period, they will have access to 3 booster session.
  Arms: Experimental: CHAMPS and mEIS

SUMMARY:
The concerning lack of research related to technology-based psychological interventions in individuals with psychosis and cannabis use disorder (CUD) led to the design a randomized control trial (RCT) with an innovative mobile health e-intervention called ICanChange (iCC). Randomized control trials (RCTs) on well-defined samples (limited to psychosis and CUD) are needed to generate evidence on e-health interventions in individuals with psychosis and CUD. As such, an RCT will be conducted to assess the acceptability and feasibility of administering this e-intervention to young people with psychosis who use cannabis. Besides having scarce cannabis interventions adapted for people with psychosis, there are other barriers to addressing problematic cannabis use, such as the challenging and inadequate access to mental health and substance use services by this population. Implementing these and other approaches in the context of a harm reduction intervention or applying other strategies seeking to minimize cannabis-related harms for people who wish to continue using cannabis may be key in helping individuals set realistic goals that are important and relevant to them.

DETAILED DESCRIPTION:
This is a multi-site, two-arm, open-label, pilot randomized control trial, involving 100 young adults diagnosed with psychosis and cannabis use disorder (CUD). Participants will be randomly assigned to either:

Arm 1. Early intervention services (EIS): early intervention for psychosis, including standard of care for psychosis and CUD following Canadian guidelines.

Arm 2. iCC + modified EIS (mEIS): The iCC is an application-based intervention that includes psychotherapeutic modules based on Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT). Participants in this arm also receive the same services as in EIS, excluding formal psychotherapeutic interventions for CUD.

Participants will complete assessments at baseline, and at 6, 12, and 24 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Young adults age 18 to 35 years old
2. Diagnosed with any psychotic disorder, which can include schizophrenia, schizoaffective disorder, bipolar disorder with psychotic features, delusional disorder, psychotic disorder not otherwise specified, brief psychotic disorder and substance-induced psychotic disorder.
3. Has been followed at an early psychosis clinic for a minimum of 3 months
4. Diagnosed with a current CUD (any severity), based on Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria
5. Currently using cannabis (used cannabis at least once in the past month)
6. Accepting an intervention for CUD to cease or decrease his/her use
7. Able to provide full informed consent
8. Available for the whole duration of the study/able to comply with study procedures
9. Able to comprehend French or English

Exclusion Criteria:

1. Any medical condition that in the opinion of the psychiatrist precludes safe participation in the study or the ability to provide fully informed consent
2. Any disabling, unstable or acute mental condition that in the opinion of the psychiatrist precludes safe participation in the study or the ability to provide fully informed consent
3. Any legal/judicial status/issue, pending legal action, or other reasons in the opinion of the study team that might prevent completion of the study
4. Presence of an additional substance use disorder that, in the opinion of the psychiatrist, precludes safe participation in the study (e.g., very unstable or severe substance use disorder)
5. Currently participating in another specific cannabis use-focused intervention (other than those which are part of the intervention and control arms)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Completion rates | Week 12
  Number of participants who completed the first section of the intervention and at least one module from section 2 related to achieving their cannabis consumption objectives or with ongoing participation in EIS.
Retention rates | Week 12
  Proportions of participants retained in the trial (completing all endpoint assessments)

SECONDARY OUTCOMES:
Acceptability (iCC usage data) | Weeks 0-24
  Number of iCC modules completed, time spent on each module, time elapsed between module initiation and completion, total time spent on iCC.
Participant satisfaction | Weeks 6, 12 & 24
  Score on the Client Satisfaction Questionnaire-I (CSQ-I). The CSQ-I is a modified version of the CSQ-8 measuring global satisfaction with a web-based intervention and and provider reports. Items are scored from 1= "does not apply to me" to 4= "Does totally apply to me". The scores for all eight items will be summed for a total score in the range 8 to 32. To calculate scores on the CSQ-I, sum item responses (range from 8-32). Higher scores indicate higher satisfaction. This collects information on the participant's satisfaction as it relates to the assigned cannabis-focused intervention.
Trial parameters | Week -4 to Week 24
  Numbers of participants who are referred, screened, eligible, consenting, randomized, initiating and completing the study
Cannabis Use | (-2-0 (baseline) and Week 6, 12 & 24
  Frequency and quantity of cannabis use in the last 14 days will be measured using the Timeline Follow Back (TLFB) which is a tool that captures self-reported drug use. The TLFB will assess the frequency of cannabis use, the self-reported days with abstinence from cannabis weekly, as well as type of cannabis products, quantity and dose/concentration in cannabinoids.

OTHER OUTCOMES:
Psychotic Symptoms | (-2-0 (baseline) and Week 6, 12 & 24
  Positive and negative symptoms of psychosis (e.g., schizophrenia) will be measured by trained staff with Positive Negative Syndrome Scale (PANSS-6) that has been recently validated in individuals with schizophrenia and shows similar psychometric properties to PANSS-30. PANSS-6 is an interviewer-administered scale, each item is scored from 1-7 based on the presence and severity of symptoms (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme). A total score of 6 reveals no psychotic symptoms and a total score of <14 is considered the cut-off for remission
Cannabis-related problems | (-2-0 (baseline) and Week 6, 12 & 24
  Cannabis-related physical, psychological, social, and functioning problems will be assessed with the Marijuana Problems Scale (MPS), which is a 19-item self-report instrument that measures change in problems related to cannabis use over time. The scale contains 19 items that represent potential negative effects of marijuana on social relationships, self-esteem, motivation and productivity, work and finances, physical health, memory impairment, and legal problems. For each item, the participant reports problems related to cannabis use in the last month by choosing one of the following three options: 0=not a problem, 1=a minor problem, 2=a serious problem. A total score is calculated, and higher scores indicate more serious problems with cannabis use.
Cannabis use frequency and abstinence | (-2-0 (baseline) and Week 6, 12 & 24
  The frequency of cannabis use (number of days in the previous 14 days weeks) and rates of point prevalence for cannabis abstinence will be assessed with the Timeline Followback (TLFB). The TLFB is a tool that captures self-reported drug use. The TLFB will assess the frequency of cannabis use, the self-reported days with abstinence from cannabis weekly, as well as type of cannabis products, quantity and dose/concentration in cannabinoids.
Other drug use | (-2-0 (baseline) and Week 6, 12 & 24
  Past two weeks other drug use according to the Timeline Follow-Back Questionnaire (TLFB) which is a tool that captures self-reported drug use in the past 14 days. The TLFB will assess the frequency of drug use, and capture self-reported days with abstinence from substance use.
Dependence severity | (-2-0 (baseline) and Week 6, 12 & 24
  Severity of cannabis dependence will be measured with the self-administered, the Severity of Dependence Scale (SDS). The SDS contains five items that measure the psychological components of dependence including control over cannabis use, anxiety over missing a dose, worry related to use, desire to stop and difficulties related to stopping using cannabis. Each item is score on a four-point scale (0=never/almost never, 1=sometimes, 2=often, 3=always/nearly always). A total score is calculated, and higher scores indicate higher levels of dependence.
Protective behaviours | (-2-0 (baseline) and Week 6, 12 & 24
  Measured with the self-administered 17-item Protective Behavioral Strategies-Marijuana (PBSM) questionnaire. The PBSM will be used to measure cannabis-related harms in the last 30 days by asking participants to rate on a six-point scale their behaviors (e.g., Avoid using before work or school) related to cannabis use (1=never, 2=rarely, 3=occasionally, 4=sometimes, 5=usually and 6=always). Mean scores will be calculated with higher scores indicating higher risk behaviors.
Confidence in resisting cannabis use | (-2-0 (baseline) and Week 6, 12 & 24
  Participant confidence in resisting cannabis use will be measured using the Drug-Taking Confidence Questionnaire (DTCQ), which is an 8-item instrument that has shown reliability and validity in measuring coping self-efficacy. Participants will rate on a 6-point scale (0= not at all confident, 20=20% confident, 40=40%, 60=60% confident, 80=80% confident; and 100=very confident) their confidence to resist cannabis use (i.e., "I would be able to resist the urge to use cannabis…" in 8 different situations e.g. "…. If other people treated me unfairly or interfered with my plans". Participant's confidence in his/her ability to resist cannabis use will be evaluated by calculating a mean score e.g., a confidence score between 0% to 20% reflects little or no confidence at all.
Life satisfaction | (-2-0 (baseline) and Week 6, 12 & 24
  The impact of psychosis and CUD on participants' life, we will be measured using the Satisfaction with Life questionnaire (SWL), which is a self-report, 18-item scale that has been validated in participants with schizophrenia and schizophrenia-related disorders. The SWL assesses individual's satisfaction with life pertaining to four domains: living situation (4 items, e.g., "How much do you like the place where you live?"), social relationships (6 items, e.g., How satisfied are you with the number of friends you have?"), work (2 items, e.g., "How satisfied are you with the kind of work that you do?") and self and present life (6 items, e.g., "How satisfied are you with yourself on the whole?"). Items are measured on a five-point Likert scale from "not at all satisfied" to "very satisfied". For each domain a mean score is calculated, and higher scores are indicative of greater satisfaction.
Healthcare utilization | (-2-0 (baseline) and Week 6, 12 & 24
  Health service utilization information including number of days of hospitalizations and number of emergency visits in the past 30 days will be collected via self-report from the participant and can be confirmed as needed through the patient medical record abstraction and contact with the case manager.
Stage of change | (-2-0 (baseline) and Week 6, 12 & 24
  To capture participants' decision stage of change related to decreasing or stopping cannabis abstinence, we will use the Precaution Adoption Model (PAPM). The PAPM consists of 7 distinct stages of health decision-making: 1) unaware of the health behavior, 2) unengaged in the decision, 3) undecided, 4) decided not to act, 5) decided to act, 6) acting and 7) maintenance. Participants will select one of 6 response options corresponding to PAPM stages 2 to 7: "At this moment, I have not thought about decreasing or stopping using cannabis", "At this moment, I am undecided about decreasing or stopping using cannabis", At this moment I do not want to decrease or stop using cannabis", "At this moment I do want to decrease or stop using cannabis", "I have recently decreased or stopped using cannabis" and "I decreased or stopped using cannabis more than one month ago".
Social support | (-2-0 (baseline)
  The availability of social support will be measured with the short form of the Social Provisions Scale (SPS-10) that consists of 2 items per dimension of support (i.e., emotional support or attachment, social integration, reassurance of worth, tangible help, orientation) for a total of 10 items. Items are measured on a four-point Likert scale from "1-totally disagree" to "4-totally agree" and a total score will be calculated. A continuous scale score is computed by summing responses to the 10 questions, with values ranging from 10 to 40. The SPS-10 summary score is not computed for respondents with data missing on any items. Higher scores can be interpreted as having higher levels of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (5):
- Canada (5):
  - Foothills Medical Centre Early Psychosis Intervention Program, Calgary, Alberta
  - Nova Scotia Early Psychosis Program, Halifax, Nova Scotia
  - Clinic Connec-T - Institut universitaire en santé mentale de Montréal, Montreal, Quebec
  - Clinique JAP, Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Clinic Notre-Dame des Victoires - Centre de Recherche CERVO, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data sharing procedure will be made developed and made available after completion of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months following the study completion.
Access Criteria: On request.

REFERENCES:
- [Derived] Tatar O, Abdel-Baki A, Wittevrongel A, Lecomte T, Copeland J, Lachance-Touchette P, Coronado-Montoya S, Cote J, Crockford D, Dubreucq S, L'Heureux S, Ouellet-Plamondon C, Roy MA, Tibbo PG, Villeneuve M, Jutras-Aswad D. Reducing Cannabis Use in Young Adults With Psychosis Using iCanChange, a Mobile Health App: Protocol for a Pilot Randomized Controlled Trial (ReCAP-iCC). JMIR Res Protoc. 2022 Nov 25;11(11):e40817. doi: 10.2196/40817. PMID 36427227